## **Official Study Title:**

The Clinical Effects of Kinesio Taping Versus Sham Taping on Pain, Kinesiophobia, Functional Mobility, and Disease Activity in Patients with Rheumatoid Arthritis: A Randomized Controlled Trial

# ClinicalTrials.gov Identifier (NCT Number):

NCT0XXXXXXX

#### **Document Date:**

30 October 2024

## **Principal Investigator:**

Ozden Baskan

Istanbul Rumeli University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation

The Effectiveness of Kinesiology Taping in Patients with Knee Rheumatoid Arthritis in Terms of Pain, Function and Kinesiophobia: A Randomised Controlled Trial

# **Background:**

## **Background:**

Rheumatoid arthritis is a chronic inflammatory disease that leads to joint pain, reduced

functional capacity, and movement-related fear. Non-pharmacological and supportive treatment methods are increasingly emphasized to improve patients' quality of life. Kinesio taping has been suggested as a potential complementary approach, but its clinical benefits compared to sham applications remain uncertain.

### **Objective:**

The aim of this study is to investigate the effects of kinesio taping compared to sham taping in patients with rheumatoid arthritis, with a particular focus on pain, functional mobility, kinesiophobia, and disease activity.

#### **Methods:**

A randomized controlled design is planned, including 30 patients with rheumatoid arthritis aged 45–65 years with moderate disease activity (DAS28: 2.6–5.1). Participants will be randomly assigned to two groups: kinesio taping or sham taping. Interventions will be applied twice a week for four weeks. Outcomes will include pain (Visual Analog Scale), disease activity (DAS28), kinesiophobia (Tampa Kinesiophobia Scale), and functional mobility (Timed Upand-Go Test). Measurements will be taken before and after the intervention period.

**Ethical Approach:** All procedures conform to the ethical standards of the Helsinki Declaration and were approved by the Istanbul Rumeli University Ethics Committee.

The Statistical analysis: The statistical evaluation of the study data will be carried out using IBM SPSS Statistics version 26.0. The distribution of quantitative variables will be examined with the Kolmogorov-Smirnov test to determine normality. Between-group comparisons of categorical variables will be performed with the Chi-square test, while continuous variables will be analyzed using the Independent Samples t-test. Pre- and post-intervention differences within each group will be assessed by the paired t-test. Statistical significance will be set at p < 0.05. In addition, effect sizes will be estimated as r values, calculated from the formula  $t / \sqrt{n}$ , in accordance with Cohen's d interpretation.